CLINICAL TRIAL: NCT01730950
Title: Randomized Phase II Trial of Concurrent Bevacizumab and Re-Irradiation Versus Bevacizumab Alone as Treatment for Recurrent Glioblastoma
Brief Title: Bevacizumab With or Without Radiation Therapy in Treating Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-1205; NCI-2012-01732 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA021661 (NIH); NCT02671981 (obsolete NCT alias)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Bevacizumab; Radiotherapy; Radiotherapy, Conformal; Proton Therapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Active Comparator): Bevacizumab every 2 weeks
  Interventions: Biological: bevacizumab
- Bevacizumab + RT (Experimental): Radiation therapy with bevacizumab every 2 weeks
  Interventions: Biological: bevacizumab; Radiation: radiation therapy

INTERVENTIONS:
Biological: bevacizumab — Staring within 14 days of randomization, IV 10mg/kg every two weeks until disease progression.
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Radiation: radiation therapy — Starting with second dose of bevacizumab, 35 Gy in 10 fractions of 3.5 Gy each delivered on consecutive treatment days (typically 5 fractions per week).
  Other Names: 3D conformal radiation therapy; photon beam radiation therapy; proton beam radiation therapy; Intensity Modulated Radiation Therapy (IMRT); Image-Guided Radiation Treatment (IGRT); 3D-CRT
  Arms: Bevacizumab + RT

SUMMARY:
This randomized phase II trial studies how well bevacizumab with or without radiation therapy works in treating patients with recurrent glioblastoma. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry cancer-killing substances to them. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. It is not yet know whether bevacizumab is more effective with or without radiation therapy in treating patients with recurrent glioblastoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish an improvement in overall survival in recurrent glioblastoma (GBM) patients receiving bevacizumab and re-irradiation compared with patients receiving bevacizumab alone.

SECONDARY OBJECTIVES:

I. To estimate and compare the rate of objective response in patients with measurable disease.

II. To estimate and compare the 6-month progression-free survival rate. III. To estimate and compare progression-free survival. IV. To estimate and compare the rate of treatment adverse events. V. To estimate and compare the rate of grade 3+ acute or delayed central nervous system (CNS) toxicity.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

In both arms, courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 1 year, every 6 months for 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of glioblastoma or variants (gliosarcoma, giant cell glioblastoma etc); patients will be eligible if the original histology was lower-grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma is made
* Patients who did not have recent surgery for their glioblastoma must have shown unequivocal radiographic evidence for tumor progression by contrast-enhanced magnetic resonance imaging (MRI) scan (or computed tomography [CT] scan for patients with non-compatible devices) CT scan within 21 days prior to registration.

  * Note: Patients who did have surgery with a post-operative contrast-enhance scan falling outside the 5 week window prior to registration, must have a repeat MRI scan (or CT scan for patients with non-compatible devices) within 21 days prior to registration.
* Patients also must have passed an interval of 6 months or greater between completion of prior radiotherapy and registration; if patients have not passed an interval of at least 6 months, they may still be eligible if they meet one or more of the following criteria:

  * New areas of tumor outside the original radiotherapy fields as determined by the investigator, or
  * Histologic confirmation of tumor through biopsy or resection, or
  * Nuclear medicine imaging, magnetic resonance (MR) spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than radiation necrosis obtained within 28 days of registration AND an interval of at least 90 days between completion of radiotherapy and registration
* Patients unable to undergo MR imaging because of non-compatible devices can be enrolled provided CT scans are obtained and are of sufficient quality; patients without non-compatible devices may not use CT scans performed to meet this requirement
* Prior history of standard dose CNS radiation of 60 Gy in 30 fractions or 59.4 Gy in 1.8 Gy fractions, or equivalent or lower doses
* Patients who have received prior treatment with non-standard radiation therapy (RT) dose and fractionation, interstitial brachytherapy, stereotactic radiosurgery, etc. are eligible
* Patients must have recovered from the toxic effects of prior therapy, and there must be a minimum time of 28 days prior to registration from the administration of any investigational agent or prior cytotoxic therapy with the following exceptions:

  * 14 days from administration of vincristine
  * 42 days from administration of nitrosoureas
  * 21 days from administration of procarbazine
* Patients having undergone recent resection of their glioblastoma (within 5 weeks prior to registration) must have recovered from the effects of surgery; for CNS related core or needle biopsies, a minimum of 7 days must have elapsed prior to registration
* Residual disease following resection of recurrent glioblastoma is not mandated for eligibility into the study; to best assess the extent of residual disease post-operatively, a post-operative or intra-operative MRI scan (or CT scan for patients with non-compatible devices) must be performed prior to registration and should be within 96 hours post surgery (although 24 hours would be optimum)
* History/physical examination, including neurologic examination, within 14 days prior to registration
* Karnofsky performance status >= 60 within 14 days prior to registration
* Complete blood count (CBC)/differential obtained within 14 days prior to registration, with adequate bone marrow function
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelets >= 75,000 cells/mm^3
* Hemoglobin >= 9.0 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin (Hgb) >= 9.0 g/dl is acceptable)
* Total bilirubin =< 2.0 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) or aspartate aminotransferase (AST) =< 2.5 times the upper limit of normal
* Serum creatinine =< 1.8 mg/dL
* Urine protein creatinine (UPC) ratio >= 1.0 within 14 days prior to registration OR urine dipstick for proteinuria >= 2+ (patients discovered to have >= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate =< 1g of protein in 24 hours to be eligible)

  * Note: UPC ratio of spot urine is an estimation of the 24-hour urine protein excretion; a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm; UPC ratio is calculated using one of the following formulas:

    * [urine protein]/[urine creatinine]: if both protein and creatinine are reported in mg/dL
    * [(urine protein) x 0.088]/[urine creatinine]: if urine creatinine is reported in mmol/L
* Patients must not be pregnant (positive pregnancy test) or breast feeding; pregnancy test must be done within 14 days prior to registration; effective contraception (men and women) must be used in patients of child-bearing potential while on trial and for 6 months after
* Patients on full-dose anticoagulants (e.g., warfarin or low molecular weight (LMW) heparin) must meet both of the following criteria:

  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
  * In-range international normalized ratio (INR) (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin, within 14 days prior to registration
* Patient must be able to provide study-specific informed consent prior to study entry

Exclusion Criteria:

* More than three relapses
* Infratentorial or leptomeningeal evidence of recurrent disease
* Recurrent or persistent tumor greater than 6 cm in maximum diameter
* Prior therapy with an inhibitor of vascular endothelial growth factor (VEGF) or VEGFR (including bevacizumab)
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1 year (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to registration
  * Transmural myocardial infarction within the last 6 months prior to registration
  * History of stroke or transient ischemic attack within 6 months prior to registration
  * Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function other than screening panel and coagulation parameters are not required for entry into this protocol
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive; protocol specific requirements may also exclude immuno-compromised patients
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Prior allergic reaction to the study drug (bevacizumab)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of a non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to registration
* Gastrointestinal bleeding or any other hemorrhage/bleeding event Common Terminology Criteria for adverse Events (CTCAE), v. 4 grade 3 or greater within 30 days prior to registration
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration (with the exception of craniotomy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Tsien, Principal Investigator — Washington University School of Medicine; Jeffrey Raizer, MD, Study Chair — Northwestern University; Adam P. Dicker, MD, PhD, Study Chair — Jefferson Medical College of Thomas Jefferson University; Martha M. Matuszak, PhD, Study Chair — University of Michigan
Locations (31):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Arizona Oncology-Deer Valley Center, Phoenix, Arizona
  - John Muir Medical Center, Walnut Creek, California
  - Yale University, New Haven, Connecticut
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Norton Health Care Pavilion - Downtown, Louisville, Kentucky
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Lowell General Hospital, Lowell, Massachusetts
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Rochester, Rochester, New York
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Summa Akron City Hospital, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Radiation Therapy Oncology Group, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Door County Cancer Center, Sturgeon Bay, Wisconsin

REFERENCES:
- [Derived] Tsien CI, Pugh SL, Dicker AP, Raizer JJ, Matuszak MM, Lallana EC, Huang J, Algan O, Deb N, Portelance L, Villano JL, Hamm JT, Oh KS, Ali AN, Kim MM, Lindhorst SM, Mehta MP. NRG Oncology/RTOG1205: A Randomized Phase II Trial of Concurrent Bevacizumab and Reirradiation Versus Bevacizumab Alone as Treatment for Recurrent Glioblastoma. J Clin Oncol. 2023 Feb 20;41(6):1285-1295. doi: 10.1200/JCO.22.00164. Epub 2022 Oct 19. PMID 36260832

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Bevacizumab (IV 10mg/kg) every 2 weeks until disease progression.
- Bevacizumab + RT: Radiation therapy (35Gy in 10 fractions of 3.5 Gy) with bevacizumab (IV 10mg/kg) every 2 weeks until disease progression.
Period: Overall Study
Arm/Group | Bevacizumab | Bevacizumab + RT
Started | 90 | 92
Eligible Population | 84 | 86
Adverse Event Population (Eligible participants who started protocol treatment) | 76 | 83
Response Population (Eligible participants with response evaluations) | 78 | 77
6-month Progression-free Analysis (Eligible participants with data at 6 months) | 79 | 81
Delayed Toxicity Population (Eligible participants on RT arm who started RT and were alive at least 91 days from the start of RT) | 0 | 83
Completed (Subjects contributing data to results are considered to have completed the study.) | 84 | 86
Not Completed | 6 | 6
Not completed — Protocol Violation | 6 | 6

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Bevacizumab + RT | Total
Number analyzed (Participants) | 84 | 86 | 170
Age, Continuous [Median (Full Range); unit: years] | 57 [25 to 87] | 60 [28 to 81] | 59 [25 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 43 | 81
  Male | 46 | 43 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 72 | 81 | 153
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 66 | 75 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 12
Karnofsky Performance Status [Count of Participants; unit: Participants] — 60 = Requires occasional assistance, but is able to care for most personal needs; 70 = Cares for self; unable to carry on normal activity or to do active work; 80 = Normal activity with effort; some signs or symptoms of disease; 90 = Able to carry on normal activity, minor signs or symptoms of disease; 100 = Normal no complaints; no evidence of disease.
  Participants
    60 | 3 | 8 | 11
    70-80 | 42 | 41 | 83
    90-100 | 39 | 37 | 76
Neurologic Function [Count of Participants; unit: Participants]
  No symptoms | 21 | 24 | 45
  Minor symptoms | 40 | 36 | 76
  Moderate symptoms (fully active) | 17 | 15 | 32
  Moderate symptoms (required assistance) | 6 | 9 | 15
  Severe symptoms | 0 | 2 | 2
Surgery for Initial Brain Tumor [Count of Participants; unit: Participants]
  Biopsy only | 8 | 7 | 15
  Subtotal resection | 20 | 25 | 45
  Gross total resection | 56 | 52 | 108
  Other | 0 | 2 | 2
Recent Resection [Count of Participants; unit: Participants]
  No / biopsy only | 49 | 57 | 106
  Yes | 35 | 29 | 64
Histologic Tumor Type [Count of Participants; unit: Participants]
  Glioblastoma (WHO Grade IV) | 79 | 82 | 161
  Gliosarcoma | 2 | 2 | 4
  Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Survival rates are estimated by the Kaplan-Meier method. The protocol specifies that the distributions of failure times will be compared between the arms, which is reported in the statistical analysis results. Eighteen-month rates are provided. Analysis was planned to occur when 135 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 52.8 months.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Bevacizumab + RT: Radiation therapy (35 Gy in 10 fractions of 3.5 Gy) with bevacizumab (IV 10mg/kg) every 2 weeks until disease progression.
Arm/Group | Bevacizumab | Bevacizumab + RT
Number analyzed (Participants) | 84 | 86
percentage of participants | 25.1 [15.2 to 35.0] | 21.6 [12.1 to 31.1]
Statistical Analysis 1: Comparison: Bevacizumab vs Bevacizumab + RT; Null hypothesis: median survival time for both arms is 9 months; alternative hypothesis: participants receiving radiation therapy plus bevacizumab will have an improvement in median survival time to 13 months. One hundred and sixty eligible participants provides 80% power to detect a 31% reduction in the hazard ratio to 0.69 at a one-sided significance level of 0.10. Analysis was planned to occur when 135 deaths were reported, expected to occur 16 to 21 months after trial closure; Test type: Superiority; p = 0.46, Log Rank; Two-side significance level = 0.05; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.70 to 1.38] — Reference level = Bevacizumab

2. Secondary Outcome: Percentage of Participants With Complete or Partial Best Response
Description: Best observed objective response determined by serial measures of the product of the two largest perpendicular cross-sectional diameters using MacDonald Criteria:
  * Complete Response (CR): complete disappearance of measurable enhancing lesion sustained ≥ 4 weeks; and no new lesions; and no corticosteroids.
  * Partial Response (PR): ≥ 50% decrease from baseline in sum of products of the measurable enhancing lesion sustained ≥ 4 weeks; and no new lesions; and stable/reduced corticosteroid dose.
  * Progression (P): ≥ 25% increase in sum of products of enhancing lesions (patient has not had steroid dose decreased since the last evaluation period); or any new lesions. A concomitant decrease in steroid dose rules out progression designation during initial 12 weeks after radiotherapy.
  * Stable Disease (SD): all of following: does not qualify for CR, PR, or P; receiving stable/decreasing doses of steroids.
  Estimated using an exact binomial distribution.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 52.8 months.
Population: Eligible participants with response evaluations
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab | Bevacizumab + RT
Number analyzed (Participants) | 78 | 77
percentage of participants | 20.5 [12.2 to 31.2] | 29.9 [20.0 to 41.4]
Statistical Analysis 1: Comparison: Bevacizumab; Test type: Superiority; p = 0.18, Chi-squared; Two-sided significance level = 0.05

3. Secondary Outcome: Percentage of Participants Progression-free at 6 Months
Description: Best observed objective response determined by serial measures of the product of the two largest perpendicular cross-sectional diameters using MacDonald Criteria:
  Progression (P): ≥ 25% increase in sum of products of enhancing lesions (patient has not had steroid dose decreased since the last evaluation period); or any new lesions. A concomitant decrease in steroid dose rules out progression designation during initial 12 weeks after radiotherapy. Progression-free at 6 months means patient alive without progression at 6 months.
Time Frame: From randomization to six months
Population: Eligible participants with data at six months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab | Bevacizumab + RT
Number analyzed (Participants) | 79 | 81
percentage of participants | 29.1 [19.4 to 40.4] | 54.3 [42.9 to 65.4]
Statistical Analysis 1: Comparison: Bevacizumab vs Bevacizumab + RT; Test type: Superiority; p = 0.001, Chi-squared; Two-sided significance level = 0.05

4. Secondary Outcome: Progression-free Survival
Description: Progression using using MacDonald Criteria is defined as ≥ 25% increase from baseline in sum of products of the two largest perpendicular cross-sectional diameters of enhancing lesions (patient has not had steroid dose decreased since the last evaluation period); or any new lesions. A concomitant decrease in steroid dose rules out progression designation during initial 12 weeks after radiotherapy. Progression-free survival time is defined as time from randomization to the date of first progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method. The protocol specifies that the distributions of failure times will be compared between the arms, which is reported in the statistical analysis results. Eighteen-month rates are provided. Analysis was planned to occur when 135 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 52.8 months.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab | Bevacizumab + RT
Number analyzed (Participants) | 84 | 86
percentage of participants | 8.9 [2.6 to 15.2] | 7.9 [1.9 to 13.9]
Statistical Analysis 1: Comparison: Bevacizumab vs Bevacizumab + RT; Test type: Superiority; p = 0.05, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.53 to 1.00] — Reference level = Bevacizumab

5. Secondary Outcome: Percentage of Participants With Grade 3+ Central Nervous System (CNS) Toxicity Within 90 Days of Start of Radiation Therapy Reported as Possibly/Probably/Definitely Related to Protocol Treatment
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 52.8 months.
Population: Eligible participants on the radiation therapy arm who started radiation therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + RT
Number analyzed (Participants) | 83
percentage of participants | 4.8 [1.3 to 11.9]

6. Secondary Outcome: Number of Participants With Grade 3+ CNS Toxicity More Than 90 Days of Start of Radiation Therapy Reported as Possibly/Probably/Definitely Related to Protocol Treatment
Description: Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. Estimated using an exact binomial distribution together with 95% confidence interval. The difference between the two groups will be tested using a chi square test.
Time Frame: From 91 days after the start of radiation therapy to end of follow-up. Maximum follow-up at the time of analysis is 58.2 months.
Population: Eligible participants on the radiation therapy arm who started radiation therapy and were alive at least 91 days from the start of radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab + RT
Number analyzed (Participants) | 83
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were to be reported every 2 months for first year, every 6 months for second year, then annually until study completion. Maximum follow-up at time of analysis was 52.8 months.
Arm/Group | Bevacizumab | Bevacizumab + RT
All-Cause Mortality (participants affected / at risk) | 4/76 | 8/83
Serious Adverse Events (participants affected / at risk) | 27/76 | 29/83
Other Adverse Events (participants affected / at risk) | 70/76 | 73/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=76) | Bevacizumab + RT (N=83)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 1 | 2
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
General disorders and administration site conditions - Other (General disorders) | 0 | 1
Neck edema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Sudden death NOS (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Investigations - Other (Investigations) | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 5 | 7
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Vasculitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=76) | Bevacizumab + RT (N=83)
Anemia (Blood and lymphatic system disorders) | 12 | 10
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 7 | 1
Blurred vision (Eye disorders) | 9 | 10
Eye disorders - Other (Eye disorders) | 5 | 7
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 12 | 8
Diarrhea (Gastrointestinal disorders) | 10 | 12
Dyspepsia (Gastrointestinal disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 20 | 14
Vomiting (Gastrointestinal disorders) | 7 | 7
Edema limbs (General disorders) | 15 | 9
Fatigue (General disorders) | 34 | 47
Gait disturbance (General disorders) | 14 | 16
General disorders and administration site conditions - Other (General disorders) | 6 | 2
Pain (General disorders) | 10 | 12
Infections and infestations - Other (Infections and infestations) | 4 | 5
Urinary tract infection (Infections and infestations) | 6 | 8
Bruising (Injury, poisoning and procedural complications) | 5 | 4
Fall (Injury, poisoning and procedural complications) | 8 | 6
Alanine aminotransferase increased (Investigations) | 7 | 11
Aspartate aminotransferase increased (Investigations) | 4 | 6
Lymphocyte count decreased (Investigations) | 11 | 7
Neutrophil count decreased (Investigations) | 8 | 4
Platelet count decreased (Investigations) | 21 | 12
Weight loss (Investigations) | 4 | 8
White blood cell decreased (Investigations) | 9 | 7
Anorexia (Metabolism and nutrition disorders) | 8 | 10
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 3
Hypokalemia (Metabolism and nutrition disorders) | 7 | 3
Hyponatremia (Metabolism and nutrition disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 9 | 5
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 8 | 5
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 6 | 5
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 4 | 5
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Ataxia (Nervous system disorders) | 4 | 2
Cognitive disturbance (Nervous system disorders) | 8 | 4
Dizziness (Nervous system disorders) | 12 | 13
Dysarthria (Nervous system disorders) | 5 | 4
Dysphasia (Nervous system disorders) | 18 | 11
Headache (Nervous system disorders) | 37 | 31
Lethargy (Nervous system disorders) | 4 | 1
Memory impairment (Nervous system disorders) | 12 | 17
Nervous system disorders - Other (Nervous system disorders) | 10 | 8
Paresthesia (Nervous system disorders) | 4 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 3
Seizure (Nervous system disorders) | 11 | 14
Anxiety (Psychiatric disorders) | 13 | 8
Confusion (Psychiatric disorders) | 11 | 12
Depression (Psychiatric disorders) | 8 | 9
Insomnia (Psychiatric disorders) | 9 | 12
Hematuria (Renal and urinary disorders) | 3 | 7
Proteinuria (Renal and urinary disorders) | 16 | 20
Renal and urinary disorders - Other (Renal and urinary disorders) | 4 | 3
Urinary incontinence (Renal and urinary disorders) | 7 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 5
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 7
Hypertension (Vascular disorders) | 33 | 29
Thromboembolic event (Vascular disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT01730950/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT01730950/ICF_001.pdf